CLINICAL TRIAL: NCT01804673
Title: Global Assessment of Treatment With IONSYS and Its Handling by Patients, Doctors and Nursing Staff in the Management of Acute Moderate to Severe Post-Surgery Pain in Hospitalised Patients
Brief Title: A Study to Evaluate the Safety and Tolerability of Fentanyl Iontophoretic Transdermal System (Fentanyl-ITS) in the Management of Post-Surgery Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was prematurely discontinued since study medication was no longer available.
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005440; FEN-PAI-3002; 2005-004087-24 (EudraCT Number)
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Fentanyl Hydrochloride; IONSYS
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl-ITS (Experimental)
  Interventions: Drug: Fentanyl-ITS

INTERVENTIONS:
Drug: Fentanyl-ITS — Fentanyl Iontophoretic Transdermal (through the skin) System (ITS) will release fentanyl at the rate of 40 microgram (mcg) (1 dose) to maximum of 240 mcg per hour (6 doses) but not more than 3.2 milligram (mg) (80 doses) per 24 hours. The duration of study treatment will be 72 hours.
  Other Names: IONSYS, Fentanyl-ITS

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the fentanyl iontophoretic transdermal (through the skin) system (fentanyl-ITS) in daily clinical practice for management of acute (a quick and severe form of illness in its early stage) moderate to severe post-operative pain (pain after surgery) including the comprehensibility and usefulness of the accompanying information material.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), single arm, and multi-center (when more than one hospital or medical school team work on a medical research study) study to evaluate safety and efficacy of the fentanyl-ITS for management of acute moderate to severe pain in post-operative participants' who have undergone elective surgery (surgery which could be postponed or not done at all without danger to the participant). The study will consists of 2 phases: screening phase (which comprises of pre-operative and post-operative stages) and an open label treatment phase. The participants will be treated with 40 microgram (mcg) of fentanyl transdermally per on-demand dose; each delivered over 10 minutes for a maximum of 6 doses (240 mcg) per hour for 24 hours and a maximum of 80 doses (3.2 milligram [mg]). Each system will inactivate at 80 doses or 24 hour, whichever occurs first. A new system will be applied every 24 hours unless the participant has used 80 doses in less than 24 hours. Maximum treatment duration of 72 hours is allowed. Participants will be expected to require parenteral (administration by injection) opioids (morphine like medications) for at least 24 hours post-operatively. This study will evaluate participant's, nurse's and physician's assessment of fentanyl-ITS under routine conditions. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with American Society of Anesthesiology (specialty concerned with the study of anesthetics [drug that is used to produce loss of pain sensation] and anesthesia [loss of sensation or feeling]) pre-operative physical status 1, 2 or 3
* Participants who are expected to remain hospitalized for at least 24 hours post-operatively (after the surgery)
* Participants, after an elective major surgical procedure (surgery which could be postponed or not done at all without danger to the participant), who are expected to have moderate or severe pain requiring parenteral (administration by injection) opioids (morphine like medications) for at least 24 hours after surgery
* Participants who are capable of understanding and cooperating with the requirements of the study and operating a transdermal (through the skin) Patients-Controlled Analgesia (PCA; methods of pain relief that may be used with or in place of analgesics [drug used to control pain])
* Participants with a pain score less than or equal to 4 (moderate pain) out of 10 on a Numerical Rating Scale (NRS), whereas 0 corresponds to no pain and 10 to the strongest imaginable pain at movement of the operated limb or body region, after titration (slow increase in drug dosage, guided by participant's responses) to comfort according to current postoperative procedures

Exclusion Criteria:

* Participants allergic or hypersensitive (very sensitive) to fentanyl or cetylpyridinium chloride or to skin adhesives
* Participants who are known or suspected to be strong opioid dependent, or who have a very high a need for strong opioids before entering the study
* Participants with a history of psychological opioid dependence before the start of the study
* Participants who are known or suspected to have abused any drug substance or alcohol in the opinion of the investigator
* Women who are pregnant, breast feeding, or planning to breast feed within 24 hrs of the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (22):
- Germany (22):
  - Augsburg
  - Berlin
  - Bremen
  - Cologne
  - Detmold
  - Dresden
  - Erfurt
  - Erlangen
  - Frankfurt
  - Halle
  - Jena
  - Kiel
  - Leipzig
  - Lünen
  - Mainz
  - Mannheim
  - Marburg
  - Münster
  - Ravensburg
  - Regensburg
  - Schwerin
  - Solingen

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl: Fentanyl Iontophoretic Transdermal (through the skin) System (ITS) releasing fentanyl at the rate of 40 microgram (mcg) (1 dose) to maximum of 240 mcg per hour (6 doses) but not more than 3.2 milligram (mg) (80 doses) per 24 hours. The duration of study treatment was up to 72 hours.
Period: Overall Study
Arm/Group | Fentanyl
Started | 174
Completed Hour 24 | 170
Completed Hour 48 | 79
Completed Hour 72 | 36
Completed | 34
Not Completed | 140
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 9
Not completed — Change to Oral Therapy | 37
Not completed — No Further Therapy Required | 84
Not completed — Use of Prohibited Medication | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Fentanyl
Number analyzed (Participants) | 174
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Global Assessment of Pain at Hour 24
Description: Participants were asked to rate their overall global assessment of pain therapy with study treatment on a 4-point verbal rating scale (poor, fair, good, excellent). Outcome of 'good' or 'excellent ' was recorded as Response while outcome of 'poor' or 'fair' was recorded as No response.
Time Frame: Hour 24
Population: Efficacy analysis set included all participants who received the study treatment at least once and who had efficacy data for the primary parameter after the 0 hour Baseline visit.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 170
percent of participants
  Response | 82.9 [76.4 to 88.3]
  No response | 17.1 [11.7 to 23.6]

2. Secondary Outcome: Number of Hours Per Day With Average Pain Intensity Less Than or Equal to 4
Description: Number of hours per day with average pain intensity less than or equal to 4 was measured on a 11-point Numeric Rating Scale (NRS) (range 0 to 10, 0=no pain; 4=mild pain; 10=strongest pain imaginable). If the participant was sleeping at time of measurement, pain intensity was assumed to be less than or equal to 4.
Time Frame: Baseline to Hour 24, Hour 24 to Hour 48 and Hour 48 to Hour 72
Population: Efficacy analysis set included all participants who received the study treatment at least once and who had efficacy data for the primary parameter after 0 hour Baseline visit. 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable for this measure at specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fentanyl
Number analyzed (Participants) | 125
hours
  Baseline to Hour 24 (n=125) | 21.3 (4.3)
  Hour 24 to Hour 48 (n= 57) | 22.2 (4.1)
  Hour 48 to Hour 72 (n= 23) | 22.7 (2.4)

3. Secondary Outcome: Change From Baseline in Pain Intensity Rating at Hour 24, 48 and 72
Description: Nursing staff asked the participants to rate their current pain intensity on 11-point NRS (range 0 to 10, 0= no pain; 10= strongest pain imaginable).
Time Frame: Baseline, Hour 24, 48 and 72
Population: Efficacy analysis set included all participants who received the study treatment at least once and who had efficacy data for primary parameter after 0 hour Baseline visit. 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable for this measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Fentanyl
Number analyzed (Participants) | 168
units on scale
  Baseline (n= 168) | 3.0 (1.2)
  Change at Hour 24 (n= 157) | -0.9 (1.7)
  Change at Hour 48 (n= 73) | -1.2 (1.8)
  Change at Hour 72 (n= 31) | -1.3 (2.1)

4. Secondary Outcome: Time Spent Out of the Bed Per Day by the Participant
Description: Participants were asked to enter the time in hours spend out of bed during the last 24 hours in the participant diary.
Time Frame: Baseline to Hour 24, Hour 24 to Hour 48 and Hour 48 to Hour 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fentanyl
Number analyzed (Participants) | 126
minutes
  Baseline to Hour 24 (n= 126) | 38.1 (94.5)
  Hour 24 to Hour 48 (n= 50) | 87.5 (121.6)
  Hour 48 to Hour 72 (n= 26) | 146.7 (193.9)

5. Secondary Outcome: Time to Mobilization
Description: Participants were asked to describe their time schedule for particular steps of mobilization by answering specific questions in the participant diary.
Time Frame: Baseline, Hours 24, 48 and 72
Population: Data was not statistically summarized but reported in individual participant listing. Due to excessive missing data it was not possible to calculate valid results for the different stages of mobilization.
Arm/Group | Fentanyl
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants With Global Assessment of Pain at Hour 48 and 72
Description: Participants were asked to give their overall global assessment of pain therapy with study treatment using a 4-point verbal rating scale (poor, fair, good, excellent). Outcome of 'good' or 'excellent ' was recorded as Response while outcome of 'poor' or 'fair' was recorded as No response.
Time Frame: Hours 48 and 72
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 79
percent of participants
  Hour 48; Response (n= 79) | 86.1 [76.5 to 92.8]
  Hour 48; No response (n= 79) | 12.7 [6.2 to 22.0]
  Hour 48; Missing (n= 79) | 1.3 [NA to NA] — Confidence Interval was not calculated for missing participants.
  Hour 72; Response (n= 36) | 97.2 [85.5 to 99.9]
  Hour 72; No response (n= 36) | 2.8 [0.1 to 14.5]

7. Secondary Outcome: Percentage of Participants With Physician Global Assessment of Pain
Description: Physicians were asked to give their overall global assessment of pain therapy with study treatment using a 4-point verbal rating scale (poor, fair, good, excellent). Outcome of 'good' or 'excellent ' was recorded as Response while outcome of 'poor' or 'fair' was recorded as No response.
Time Frame: Hours 24, 48 and 72
Population: Efficacy analysis set included all participants who received the study treatment at least once and who had efficacy data for primary parameter after 0 hour Baseline visit. 'n' signifies those participants evaluable for this measure at the specified time point.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 170
percent of participants
  Hour 24; Response (n= 170) | 88.2 [82.4 to 92.7]
  Hour 24; No response (n= 170) | 11.2 [6.9 to 16.9]
  Hour 24; Missing (n= 170) | 0.6 [NA to NA] — Confidence Interval was not calculated for missing participants.
  Hour 48; Response (n= 79) | 88.6 [79.5 to 94.7]
  Hour 48; No response (n= 79) | 11.4 [5.3 to 20.5]
  Hour 72; Response (n= 36) | 97.2 [85.5 to 99.9]
  Hour 72; No response (n= 36) | 2.8 [0.1 to 14.5]

8. Secondary Outcome: Percentage of Participants With Nursing Staff Global Assessment of Pain
Description: Nursing Staff were asked to give their overall global assessment of pain therapy with study treatment using a 4-point verbal rating scale (poor, fair, good, excellent). Outcome of 'good' or 'excellent ' was recorded as Response while outcome of 'poor' or 'fair' was recorded as No response.
Time Frame: Hours 24, 48 and 72
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 170
percent of participants
  Hour 24; Response (n= 170) | 87.1 [81.1 to 91.7]
  Hour 24; No response (n= 170) | 12.4 [7.8 to 18.3]
  Hour 24; Missing (n= 170) | 0.6 [NA to NA] — Confidence Interval was not calculated for missing participants.
  Hour 48; Response (n= 79) | 88.6 [79.5 to 94.7]
  Hour 48; No response (n= 79) | 11.4 [5.3 to 20.5]
  Hour 72; Response (n= 36) | 97.2 [85.5 to 99.9]
  Hour 72; Missing (n= 36) | 2.8 [NA to NA] — Confidence Interval was not calculated for missing participants.

9. Secondary Outcome: Physician's Evaluation of Participant's Ability to Undergo Physiotherapy or Mobilization
Description: Physicians were asked to rate the participant's ability to undergo physiotherapy or mobilization by responding to following questions of a questionnaire: Part 1 A- Does the surgical procedure performed allow the mobilization of the participant, C- Was the mobilization of the participant limited due to pain, D- Is the participant in a condition to undergo physiotherapy; Part 2 A- Was it possible to mobilize the participant sooner than with other pain therapies, B- Does the participant move more, C- Is the participant less afraid of moving. For Part 1-Question C, 'Partial' indicates that mobilization of participant was moderately limited due to pain.
Time Frame: Hours 24, 48 and 72
Population: Efficacy analysis set included all participants who received the study treatmentat least once and who had efficacy data for primary parameter after 0 hour Baseline visit. 'n' signifies participants evaluable at specified time point for specified item.
Measure: Number; unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 170
percent of participants
  Hour 24 Part 1-Question A; Yes (n=170) | 95.3
  Hour 24 Part 1-Question A; No (n=170) | 4.7
  Hour 24 Part 1-Question C; Yes (n=170) | 16.5
  Hour 24 Part 1-Question C; No (n=170) | 39.4
  Hour 24 Part 1-Question C; Partial (n=170) | 43.5
  Hour 24 Part 1-Question C; Missing (n=170) | 0.6
  Hour 24 Part 1-Question D; Yes (n=170) | 91.8
  Hour 24 Part 1-Question D; No (n=170) | 8.2
  Hour 24 Part 2-Question A; Yes (n=170) | 30.6
  Hour 24 Part 2-Question A; No (n=170) | 62.4
  Hour 24 Part 2-Question A; Missing (n=170) | 7.1
  Hour 24 Part 2-Question B; Yes (n=170) | 54.1
  Hour 24 Part 2-Question B; No (n=170) | 44.7
  Hour 24 Part 2-Question B; Missing (n=170) | 1.2
  Hour 24 Part 2-Question C; Yes (n=170) | 58.8
  Hour 24 Part 2-Question C; No (n=170) | 41.2
  Hour 48 Part 1-Question A; Yes (n=79) | 92.4
  Hour 48 Part 1-Question A; No (n=79) | 2.5
  Hour 48 Part 1-Question A; Missing (n=79) | 5.1
  Hour 48 Part 1-Question C; Yes (n=79) | 8.9
  Hour 48 Part 1-Question C; No (n=79) | 51.9
  Hour 48 Part 1-Question C; Partial (n=79) | 32.9
  Hour 48 Part 1-Question C; Missing (n=79) | 6.3
  Hour 48 Part 1-Question D; Yes (n=79) | 88.6
  Hour 48 Part 1-Question D; No (n=79) | 6.3
  Hour 48 Part 1-Question D; Missing (n=79) | 5.1
  Hour 48 Part 2-Question A; Yes (n=79) | 40.5
  Hour 48 Part 2-Question A; No (n=79) | 53.2
  Hour 48 Part 2-Question A; Missing (n=79) | 6.3
  Hour 48 Part 2-Question B; Yes (n=79) | 68.4
  Hour 48 Part 2-Question B; No (n=79) | 25.3
  Hour 48 Part 2-Question B; Missing (n=79) | 6.3
  Hour 48 Part 2-Question C; Yes (n=79) | 63.3
  Hour 48 Part 2-Question C; No (n=79) | 31.6
  Hour 48 Part 2-Question C; Missing (n=79) | 5.1
  Hour 72 Part 1-Question A; Yes (n=36) | 91.7
  Hour 72 Part 1-Question A; Missing (n=36) | 8.3
  Hour 72 Part 1-Question C; Yes (n=36) | 5.6
  Hour 72 Part 1-Question C; No (n=36) | 52.8
  Hour 72 Part 1-Question C; Partial (n=36) | 30.6
  Hour 72 Part 1-Question C; Missing (n=36) | 11.1
  Hour 72 Part 1-Question D; Yes (n=36) | 86.1
  Hour 72 Part 1-Question D; No (n=36) | 2.8
  Hour 72 Part 1-Question D; Missing (n=36) | 11.1
  Hour 72 Part 2-Question A; Yes (n=36) | 41.7
  Hour 72 Part 2-Question A; No (n=36) | 47.2
  Hour 72 Part 2-Question A; Missing (n=36) | 11.1
  Hour 72 Part 2-Question B; Yes (n=36) | 58.3
  Hour 72 Part 2-Question B; No (n=36) | 30.6
  Hour 72 Part 2-Question B; Missing (n=36) | 11.1
  Hour 72 Part 2-Question C; Yes (n=36) | 61.1
  Hour 72 Part 2-Question C; No (n=36) | 27.8
  Hour 72 Part 2-Question C; Missing (n=36) | 11.1

10. Secondary Outcome: Comprehensibility of the Information Material (IM): Physician Questionnaire Responses
Description: Physicians were asked to evaluate the IM for fentanyl-ITS (IONSYS) by responding to following questions of a questionnaire: Part2 D- Would you use IONSYS again, E- Would you prefer IONSYS to intravenous patient controlled analgesia (IV PCA); Part3 A- Was IM easy to understand, B- Did IM help you to use system properly.
Time Frame: Hour 72
Population: Efficacy analysis set included all participants who received the study treatment at least once and who had efficacy data for primary parameter after 0 hour Baseline visit. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 36
percent of participants
  Part 2-Question D; Yes | 83.3
  Part 2-Question D; No | 5.6
  Part 2-Question D; Missing | 11.1
  Part 2-Question E; Yes | 77.8
  Part 2-Question E; No | 11.1
  Part 2-Question E; Missing | 11.1
  Part 3-Question A; Yes | 88.9
  Part 3-Question A; Missing | 11.1
  Part 3-Question B; Yes | 88.9
  Part 3-Question B; Missing | 11.1

11. Secondary Outcome: Comprehensibility of the Information Material (IM): Nursing Staff Questionnaire Responses
Description: Nursing staff were asked to evaluate the IM for IONSYS by responding to following questions of a questionnaire: IM A- Was IM easy to understand, B- Did IM help you to use system properly; IONSYS PCA A- Is system easy to handle, B- Did participant need help in using system, C- Do you feel confident using IONSYS; IV PCA- Are you experienced in using IV PCA; IONSYS PCA D- Could participant get mobilized sooner, E- Does participant move more, F- Is participant less afraid of moving, G- Were hospital logistics for IONSYS easier to handle.
Time Frame: Hour 72
Population: Efficacy analysis set included all participants who received the study treatment at least once and who had efficacy data for primary parameter after 0 hour Baseline visit.
Measure: Number; unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 170
percent of participants
  IM-Question A; Yes | 97.1
  IM-Question A; Missing | 2.9
  IM-Question B; Yes | 95.9
  IM-Question B; No | 1.2
  IM-Question B; Missing | 2.9
  IONSYS PCA-Question A; Yes | 95.3
  IONSYS PCA-Question A; No | 1.8
  IONSYS PCA-Question A; Missing | 2.9
  IONSYS PCA-Question B; Yes | 23.5
  IONSYS PCA-Question B; No | 73.5
  IONSYS PCA-Question B; Missing | 2.9
  IONSYS PCA-Question C; Yes | 90.0
  IONSYS PCA-Question C; No | 5.9
  IONSYS PCA-Question C; Missing | 4.1
  IV PCA-Question; Yes | 84.1
  IV PCA-Question; No | 10.6
  IV PCA-Question; Missing | 5.3
  IONSYS PCA-Question D; Yes | 31.2
  IONSYS PCA-Question D; No | 48.8
  IONSYS PCA-Question D; Missing | 20.0
  IONSYS PCA-Question E; Yes | 52.9
  IONSYS PCA-Question E; No | 32.4
  IONSYS PCA-Question E; Missing | 14.7
  IONSYS PCA-Question F; Yes | 47.6
  IONSYS PCA-Question F; No | 37.6
  IONSYS PCA-Question F; Missing | 14.7
  IONSYS PCA-Question G; Yes | 71.8
  IONSYS PCA-Question G; No | 12.4
  IONSYS PCA-Question G; Missing | 15.9

12. Secondary Outcome: Comprehensibility of the Information Material (IM): Participant Questionnaire Responses
Description: Participants were asked to evaluate the IM for IONSYS by responding to following questions of a questionnaire: A- Is IONSYS easy to use, B- Were you able to operate the system by yourself after receiving instructions, C- Have you found button yourself, D- Was pressing button easy, E- Have you heard system's beeps, F- Was IONSYS IM easy to understand, G- Did IM help you to use system, H- Did you have problems falling asleep, I- Could you move easily in bed, J- Did system bother you during physiotherapy, K- Do you perceive use of such system as modern treatment standard.
Time Frame: Hour 72
Population: as for outcome 11
Measure: Number; unit: percent of participants
Arm/Group | Fentanyl
Number analyzed (Participants) | 170
percent of participants
  Question A; Yes | 77.1
  Question A; No | 1.2
  Question A; Missing | 21.8
  Question B; Yes | 77.6
  Question B; No | 1.2
  Question B; Missing | 21.2
  Question C; Yes | 78.8
  Question C; Missing | 21.2
  Question D; Yes | 77.6
  Question D; No | 1.2
  Question D; Missing | 21.2
  Question E; Yes | 72.9
  Question E; No | 4.7
  Question E; Missing | 22.4
  Question F; Yes | 75.9
  Question F; No | 1.8
  QuestionF; Missing | 22.4
  Question G; Yes | 75.9
  Question G; No | 0.6
  Question G; Missing | 23.5
  Question H; Yes | 30.0
  Question H; No | 46.5
  Question H; Missing | 23.5
  Question I; Yes | 60.6
  Question I; No | 17.1
  Question I; Missing | 22.4
  Question J; Yes | 4.1
  Question J; No | 71.2
  Question J; Missing | 24.7
  Question K; Yes | 75.3
  Question K; No | 1.8
  Question K; Missing | 22.9

13. Secondary Outcome: Post-Operative Phase (PPP33) Quality of Life Questionnaire Score
Description: The PPP33 questionnaire has an overall score and 8 subscales that represent different aspects of the post-operative quality of life: information, autonomy, communication, physical complaints, pain, rest, fear and accommodation. Answers to individual question are scored with values 1 to 4. Summary scores are calculated by adding values for each question. Subscores ranges depend on the number of questions evaluated (2 to 7 questions). The overall score ranges from 1 to 100. Higher scores indicate less pain.
Time Frame: Hour 72
Population: Efficacy analysis set included all participants who received the study treatment at least once and who had efficacy data for the primary parameter after the 0 hour Baseline visit. 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Fentanyl
Number analyzed (Participants) | 105
units on scale | 76.8 (9.4)

ADVERSE EVENTS:
Time Frame: From signing of informed consent until Day 7 after end of treatment
Description: Treatment-emergent are events between first dose of study drug and up to 7 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Arm/Group | Fentanyl
Serious Adverse Events (participants affected / at risk) | 3/174
Other Adverse Events (participants affected / at risk) | 86/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (N=174)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1
Impaired healing (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (N=174)
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 16
Flatulence (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Application site erythema (General disorders) | 18
Application site vesicles (General disorders) | 5
Application site burn (General disorders) | 4
Application site irritation (General disorders) | 3
Application site pruritus (General disorders) | 3
Application site oedema (General disorders) | 2
Application site pain (General disorders) | 2
Dizziness (Nervous system disorders) | 6
Hypotension (Vascular disorders) | 6
Procedural nausea (Injury, poisoning and procedural complications) | 4
Procedural vomiting (Injury, poisoning and procedural complications) | 4
Erythema (Skin and subcutaneous tissue disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2
Oxygen saturation decreased (Investigations) | 2
Sleep disorder (Psychiatric disorders) | 2

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued after enrolling 184 of 200 planned participants because the study medication was no longer available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No